CLINICAL TRIAL: NCT06465069
Title: A Phase 1a/1b Study of LY4052031, an Antibody-Drug Conjugate Targeting Nectin-4, in Participants With Advanced or Metastatic Urothelial Carcinoma or Other Solid Tumors
Brief Title: A Study of LY4052031 in Participants With Advanced or Metastatic Urothelial Cancer or Other Solid Tumors
Acronym: NEXUS-01
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18882; 2024-512927-36-00 (EU CTIS Number); J5I-OX-JZYA (Other: Eli Lilly and Company); LOXO-LNC-24001 (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Solid Tumor; Recurrent Solid Tumor; Advanced Solid Tumor; Urinary Bladder Neoplasm; Triple Negative Breast Cancer; Non-small Cell Lung Cancer; Esophageal Cancer; Pancreatic Cancer; Ovarian Cancer; Cervical Cancer; Head and Neck Squamous Cell Carcinoma; Prostate Cancer; Renal Pelvis Cancer; Bladder Cancer
Keywords: Bladder Cancer; Bladder Neoplasm; Bladder Urothelial Carcinoma; Urinary Bladder Cancer; Urinary Tract Cancer; Urothelial Neoplasms; Renal Pelvis Cancer; Ureter Cancer; Nectin-4; Antibody Drug Conjugate (ADC); Triple Negative Breast Cancer (TNBC); Non-small Cell Lung Cancer (NSCLC); Head and Neck Squamous Cell Carcinoma (HNSCC)
MeSH Terms: conditions — Neoplasm Metastasis; Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Esophageal Neoplasms; Pancreatic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms; Squamous Cell Carcinoma of Head and Neck; Prostatic Neoplasms; Urologic Neoplasms; Ureteral Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LY4052031 (Dose-escalation, Cohort A1) (Experimental): Escalating doses of LY4052031 administered intravenously (IV).
  Interventions: Drug: LY4052031
- LY4052031 (Dose-optimization, Cohort A2) (Experimental): Comparing 2 or more doses (evaluated during dose escalation) of LY4052031 administered IV.
  Interventions: Drug: LY4052031
- LY4052031 (Dose-expansion, Cohort B1, B2, C1) (Experimental): LY4052031 administered IV.
  Interventions: Drug: LY4052031

INTERVENTIONS:
Drug: LY4052031 — Intravenous

SUMMARY:
The purpose of this study is to find out whether the study drug, LY4052031, is safe, tolerable and effective in participants with advanced, or metastatic solid tumors including urothelial cancer. The study is conducted in two parts - phase Ia (dose-escalation, dose-optimization) and phase Ib (dose-expansion). The study will last up to approximately 4 years.

DETAILED DESCRIPTION:
This is a Phase 1a/1b multicenter, open-label study in participants with advanced or metastatic solid tumor malignancies known to express Nectin 4. This study evaluates an antibody-drug conjugate that binds to the protein nectin-4, which is expressed on certain cancer cells, delivering the drug to the cancer. This study is comprised of two phases: Dose Escalation and Dose Optimization (1a), and Dose expansion (1b). Phase 1a will assess the safety, tolerability, and pharmacokinetics of LY4052031 to determine the recommended phase 2 dose (RP2D)/optimal dose. Phase 1b will evaluate efficacy and safety of LY4052031 at the RP2D/optimal dose in expansion cohorts based on tumor type and/or treatment history.

ELIGIBILITY:
Inclusion Criteria:

* Have one of the following solid tumor cancers:

  * Cohort A1: urothelial carcinoma, triple negative breast cancer, non-small cell lung cancer, esophageal cancer, pancreatic cancer, ovarian cancer, cervical cancer (squamous cell carcinoma), head and neck squamous cell carcinoma or prostate cancer
  * Cohort A2/B1/B2: urothelial carcinoma
  * Cohort C: triple negative breast cancer, non-small cell lung cancer, ovarian cancer, cervical cancer, HNSCC (head and neck squamous cell carcinoma), esophageal cancer, pancreatic cancer, or prostate cancer
* Prior Systemic Therapy Criteria:

  * Cohort A1/C: Individual has received all standard therapies for which the participant was deemed to be an appropriate candidate by the treating investigator; OR there is no standard therapy available for the disease. There is no restriction on number of prior therapies
  * Cohort A2/B1/B2: Individual must have received at least one prior regimen in the advanced or metastatic setting. There is no restriction on number of prior therapies.
* Prior enfortumab vedotin specific requirements:

  * Cohorts A1/A2/C: prior treatment with enfortumab vedotin is allowed, but not required
  * Cohort B1: individual must be enfortumab vedotin naive in the advanced/metastatic setting
  * Cohort B2: individual must have received enfortumab vedotin in the metastatic/advanced setting.
* Measurability of disease

  * Cohort A1: measurable or non-measurable disease as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST 1.1)
  * Measurable disease is required as defined by Response Evaluation Criteria in Solid Tumors v1.1 (RECIST v1.1) for all Cohorts. Cohort A1 may permit non-measurable disease as defined by RECIST v1.1
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Have adequate archival tumor tissue sample available or undergo a screening biopsy if allowed per country specific regulations

Exclusion Criteria:

* Individual with known or suspected uncontrolled CNS metastases
* Individual with uncontrolled hypercalcemia
* Individual with uncontrolled diabetes
* Individual with evidence of corneal keratopathy or keratitis, and history of corneal transplant
* Any serious unresolved toxicities from prior therapy
* Significant cardiovascular disease
* Recent thromboembolic event and/or clinically significant bleeding disorder
* Prolongation of QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms
* History of pneumonitis/interstitial lung disease
* History of Grade ≥3 skin toxicity when receiving enfortumab vedotin
* Individuals who are pregnant, breastfeeding or plan to breastfeed during study or within 30 days of last dose of study intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: To determine the recommended phase 2 dose (RP2D) optimal dose(s) of LY4052031 | Cycle 1 (21 Days)
  Number of participants with dose-limiting toxicities (DLTs)
Phase 1b: To assess the antitumor activity of LY4052031 Monotherapy: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) properties of LY4052031: Minimum Plasma Concentration (Cmin) | Cycle 1 (21 Days)
  PK: Cmin of LY4052031
To characterize the PK properties of LY4052031: Area under the concentration versus time curve (AUC) | Cycle 1 (21 Days)
  PK: AUC of LY4052031
To evaluate the preliminary antitumor activity of LY4052031: Overall response rate (ORR) | Up to Approximately 48 Months or 4 Years
  ORR per investigator assessed Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1))
To evaluate the preliminary antitumor activity of LY4052031: Duration of response (DOR) | Up to Approximately 48 Months or 4 Years
  DOR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4052031: Time to response (TTR) | Up to Approximately 48 Months or 4 Years
  TTR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4052031: Progression free survival (PFS) | Up to Approximately 48 Months or 4 Years
  PFS per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4052031: Disease control rate (DCR) | Up to Approximately 48 Months or 4 Years
  DCR per investigator assessed RECIST 1.1
To evaluate the preliminary antitumor activity of LY4052031: Overall survival (OS) | Up to Approximately 48 Months or 4 Years
  OS per investigator assessed RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (28):
- United States (15):
  - City of Hope National Medical Center, Duarte, California
  - Sarah Cannon Research Institute at HealthOne, Denver, Colorado
  - Florida Cancer Specialists and Research Institute, St. Petersburg, Florida
  - University of Chicago Hospital, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest Cancer and Hematology Centers of W Michigan, Grand Rapids, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - START Mountain Region, West Valley City, Utah
- Australia (2):
  - St Vincent's Hospital, Darlinghurst
  - Linear Clinical Research, Nedlands
- Institut Gustave Roussy (Igr), Villejuif, France
- Japan (3):
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - The Cancer Institute Hospital of JFCR, Kōtō City
  - Aichi Cancer Center Hospital, Nagoya
- Asan Medical Center, Seoul, South Korea
- Spain (4):
  - Catalan Institute of Oncology Duran i Reynals Hospital, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Madrid Norte Sanchinarro, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
- United Kingdom (2):
  - St Bartholomew's Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study of LY4052031 in Participants With Advanced or Metastatic Urothelial Cancer or Other Solid Tumors — https://trials.lilly.com/en-US/trial/503555